CLINICAL TRIAL: NCT04248270
Title: A Noval Tau Tracer ([18F]PM-PBB3) in Young Onset Dementia: Clinical and Neuroimaging Study
Brief Title: A Noval Tau Tracer in Young Onset Dementia
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Hsu, Jung-Lung, MD, Associate Professor, Chang Gung Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201802151A0
Record Dates: First submitted 2020-01-21; First posted 2020-01-30 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Alzheimer's Disease; Vascular Dementia; Dementia
MeSH Terms: conditions — Alzheimer Disease; Dementia, Vascular; Dementia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The relationship between image and AD disease (Other): To evaluate the relationship between F-18-PMPBB3 PET image uptake pattern and AD disease classifications.
  Interventions: Drug: 18F-PM-PBB3

INTERVENTIONS:
Drug: 18F-PM-PBB3 — All scans will be acquired in pairs of 18F-florbetapir(18F-AV45) and/or18F-PM-PBB3 PET scans (if patient select), performed on separate days, and at least 2 days apart, with either scan performed first. The 18F-florbetapir and 18F-PM-PBB3 protocol will entail the inon of 5±2mCi of tracer followed by an uptake phase of 50 min during which time the state of the subject is not important. After 40 minutes, subjects will be positioned and 4 x 5 min frames of emission data will be collected right at 50 min after tracer injection. PET/MRI scans will precede this acquisition with a MRI scan for attenuation correction; PET-only scanners will perform a transmission scan following the emission scan.

SUMMARY:
Dementia is a clinical syndrome which characterized by progressive cognitive impairment, behavior disturbance and dysfunction of daily activity. In aging population, Alzheimer's dementia (AD) is the most common late onset dementia which occupied about 50-75%, the vascular dementia, frontotemporal lobardegeneration (FTLD) and corticobasal syndrome is followed. On the other hand, the young onset dementia (YOD), which represents the onset of dementia before65 years old, is only about 1/10 to 1/100 proportion of late onset dementia. The YOD is different from late onset dementia in the proportion of degenerative subtype (e.g. the FTLD is more frequent than AD). Besides, frequent atypical presentation of clinical syndrome in the YOD which characterize the different variant of AD made the early accurate diagnosis of AD is more difficult. Currently, there is no available data to describe the proportion of subtype in YOD in Taiwan. In AD dementia, two important biomarkers are amylod plaque made by ß-amyloid protein and neurofibrillary tangle made by phosphorylation tau protein. In the past, they only can be seen under the microscope findings at autopsy study. Recently, the new amyloid tracer and tau tracer had been developed and could evaluate the deposition of amyloid and tau protein in human brain. These progresses had substantially improved the accurate diagnosis of degenerative dementia. A noval tau tracer [ 18F]PM-PBB3, which had substantially improved the off-target binding and more clear background in human brain than previous tau tracer. In current project, investigator will aim to consecutive collect 50 YOD due to the neurodegeneration in 3 years using the NIA-AA research framework system(ATN system) to achieve accurate diagnosis of the dementia subtype by the detail clinical neurology study, neuropsychological examination, amyloid positron emission tomography (PET) and tau PET study. In the first year, investigator will perform feasibility study to explore the topographical tau distribution in different subtype of YOD. In the next 2 years, investigator will perform a large scale study in a group of YOD to understand the amyloid and tau deposition and their association with clinical parameters. From current project, investigator could understand the tau deposition in different YOD subtype. Investigator also could understand the correlation between clinical phenotype and molecular pathology. Investigator will use a mathematic model to construct the model of diffusion kurtosis imaging from brain magnetic resonance imaging (MRI) and relate the white matter integrity with amyloid and tau PET imaging.

ELIGIBILITY:
Inclusion Criteria Subjects

Very mild to moderate stage YOD inclusion criteria:

Age between 20-75 years old.

YOD is defined by the dementia onset before age 65 years old. The dementia syndrome is based on the NIA-AA criteria of all-cause of dementia . Briefly it required:

1. Interfere with the ability to function at work or at usual activities.
2. Represent a decline from previous levels of functioning and performing.
3. Cognitive impairment is detected and diagnosed through a combination of a). history-taking form the patient and a knowledgeable informant b). an objective cognitive assessment, either a 'bedside' mental status examination or neuropsychological testing.
4. The cognitive or behavioral impairment involves a minimum of two of the below domains: impaired ability to acquire and remember new information, impaired reasoning and handling of complex tasks poor judgment, impaired visuospatial abilities, impaired language functions, changes in personality, behavior or comportment symptoms.

The severity of dementia is limited from very mild to moderate stage in current project. The definition of very mild to moderate stage of dementia is based on the clinical dementia rating scale (CDR) from 0.5-2 YOD_2019 3 Exclusion Criteria

1. Implantation of metal devices including cardiac pacemaker, intravascular metal devices.
2. Major systemic diseases including coronary arterial disease, heart failure, uremia, hepatic failure, prominent strokes, acute myocardial infarction, poorly controlled diabetes, previous severe head injury, intracranial operation, hypoxia, sepsis or severe infectious diseases.
3. Major psychiatric disorders, drug or alcohol abuse and major depression
4. Pregnant women or breast- feeding women.
5. Patients in whom MRI was contraindicated or patient had claustrophobia.
6. History of severe allergic or anaphylactic reactions particularly to the tested drugs.
7. History of positive test for human immunodeficiency virus (HIV).
8. Indication of impaired liver function as shown by an abnormal liver function profile at screening (eg. repeated values of aspartate aminotransferase [AST] and alanine aminotransferase [ALT] ≧ 3X the upper limit of normal values).

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-02-20 (Estimated); Primary Completion 2023-08-17 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
understand the proportion of subtype in YOD | 3 years
  investigator would be able to understand the proportion of subtype in YOD
understand the mean tau deposition in different region of interest from subtype of YOD | 3 years
  investigator will perform image analysis to understand tau deposition in different subtype of YOD based on 18F-PM-PBB3 tau tracer image. The mean intensity from selected region of interest will be recorded for different group comparison.
understand the mean tau intensity in different region of interest and find correlation with cognition | 3 years
  investigator will perform association study to explore clinical measurements such as cognition and demographic data associate with tau intensity from different region of interest